CLINICAL TRIAL: NCT05069142
Title: A Study Evaluating the Feasibility of a Peri-Operative Rehabilitation Program for Inguinal Hernia Repair Surgery to Reduce Risk of Post-Surgical Pain
Brief Title: Peri-Operative Rehab Program for Inguinal Hernia Repair Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00106451
Record Dates: First submitted 2021-09-22; First posted 2021-10-06 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Inguinal Hernia
Keywords: rehabilitation; prehabilitation
MeSH Terms: conditions — Hernia, Inguinal | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Pilot Parallel-Group Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Assessors are blind to group status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 15 participants will be randomly selected to the intervention group. These individuals will receive six weeks of pre-operative exercise instruction and education, as well as six weeks of graduated post-operative exercise instruction, beginning at three weeks post-op with the surgeons clearance.
  Interventions: Other: Rehabilitation
- Control group (No Intervention): 15 participants will be randomly selected to the control group. This group will receive pre-operative education in the form of videos regarding the procedure and pain. They will not receive exercise instruction.

INTERVENTIONS:
Other: Rehabilitation — Pre- and post-operative exercise and education.
  Arms: Intervention group

SUMMARY:
Inguinal hernia repair is one of the most common surgeries, with more than 20 million performed globally each year. It is estimated that approximately 15% of patients undergoing inguinal hernia repair will experience persistent post-surgical pain that could last months to years. Evidence from related procedures indicates that better surgical preparation through pre-operative exercise and education (i.e. Prehabilitation) followed by ongoing post-surgical rehabilitation leads to more rapid recovery, return to activities and lower likelihood of persistent post-surgical pain. The investigators will determine the feasibility of a peri-operative rehabilitation program (pre- and post-surgery) and our study protocol for patients undergoing inguinal hernia repair surgery. The investigators hypothesize that: 1) our peri-operative intervention will be feasible and safe to undertake within a clinical setting; 2) adequate numbers will be enrolled to justify a larger trial; and that 3) our outcome measurement protocol will provide meaningful information with high response rate and low attrition after 3 months.

DETAILED DESCRIPTION:
Inguinal hernia repair is one of the most common surgeries performed globally, with more than 20 million performed each year. Not only does this huge number of surgeries have a substantial direct economic burden on healthcare systems, there is also indirect impact from time off work and decreased productivity due ongoing post-surgical pain requiring extended time spent on modified duties. It is estimated that approximately 15% of patients undergoing inguinal hernia repair will experience persistent post-surgical pain that could last months to years. Furthermore, current clinical guidelines for return to work and activity after inguinal hernia repair are inconsistently informed by evidence, highly variable, and outdated. Forbes et al (2012) found that the average patient undergoing inguinal hernia repair experiences more than 40 days of short-term disability despite indications that earlier return to activity is safe (i.e. will not lead to repair failure) and likely beneficial for reducing chronic pain and disability.

Evidence from related procedures indicates that better surgical preparation through pre-operative exercise and education (i.e. Prehabilitation) followed by ongoing post-surgical rehabilitation leads to more rapid recovery, return to activities and lower likelihood of persistent post-surgical pain. Prehabilitation was first described in the 1940's when the British Army developed a prehabilitation program as part of an experiment to increase the quality of recruits. The concept of prehabilitation gained traction within the medical community when Topp et. al. and Ditmyer et. al. promoted a theoretical model of prehabilitation, positing that patients who participate in presurgical exercise with the goal of improving functional capacity may experience more rapid postoperative recovery than patients who remain physically inactive through the preoperative period. Prehab has also been shown to increase self-efficacy, a moderator of pain catastrophizing and fear avoidance beliefs, that are important factors linked to the pain experience of those with persistent pain. The investigators propose that this theoretical model can be extrapolated to inguinal hernia repair and theorize that prehabilitation will increase patients' preoperative self-efficacy, allowing them to more rapidly regain abilities, subsequently shortening duration of modified duties and decreasing likelihood of persistent post-surgical pain.

Little information is available regarding the use of prehabilitation in the context of inguinal hernia repair. There have been numerous studies looking at prehabilitation in orthopedics, cardiovascular surgery, and prior to major abdominal surgeries, but limited studies for inguinal hernia repair. A randomized control study by Liang et. al. examined the impact of prehabilitation on ventral hernia recurrence and post-operative complications. They concluded that patients undergoing prehabilitation have a higher likelihood of being hernia-free and complication-free 30 days postoperatively. Notably, this study is limited in that only obese patients were included, and outcomes only included recurrence and complications. No studies were located examining the impact of prehabilitation on recovery time, post-surgical pain, and return to activity after inguinal hernia repair. However psychosocial factors such as pain catastrophizing appear to be important predictors. Typical practice guidelines often recommend limiting activity for at least 3 months to avoid re-rupture. However, these guidelines are based on expert opinion due to a lack of quality research and can pose a risk in building unhelpful beliefs about pain, fear of movement and poor coping strategies. Research is needed to inform practice guidelines and return-to-activity recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo first-time inguinal hernia repair surgery after a physical examination identified signs and symptoms consistent with inguinal hernia (direct or indirect hernia)
* Willingness to participate in a targeted peri-operative exercise program
* 18+ years of age
* No medical contraindications to participation in exercise
* Employed full-time and required to lift at least 10kg for work

Exclusion Criteria:

* Previous inguinal hernia
* Body Mass Index >35 since morbidly obese patients experience more surgical complications
* Specific contra-indications that will be screened for include associated medical conditions that preclude exercise, this includes uncontrolled medical conditions including diabetes, hypertension, vertigo, congestive heart failure, chronic obstructive pulmonary disease, intra-abdominal ascites, or pre-existing malnutrition. We will also screen for use or narcotics, bone and joint conditions of the spine or extremities, or history of other abdominal surgeries.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Pain Scale | 3 Months after the operation
  Post-surgical pain intensity ratings will be measured on a 0-100mm Visual Analogue Scale, a valid measure of pain intensity.

SECONDARY OUTCOMES:
Carolinas Comfort Scale (CCS) | 3 Months after the operation
  Post-surgical pain quality will be measured using the Carolinas Comfort Scale (CCS), a questionnaire for evaluating pain and sensations experienced by patients after inguinal hernia operations.
Change in scores on the Short-Form Functional Capacity Evaluation | Changes between baseline to three months after the operation.
  The Short-Form Functional Capacity Evaluation is a performance-based test of work function. In this test, patients are tested on 5 key activities of work performance (lifting, standing, trunk rotation, crouching, forward trunk flexion). Performance on each scale is compared to required job demands and the number of "failed" items is summed (0 to 5 failures). Short-Form Functional Capacity Evaluation is a valid indicator of work ability that has been found predictive of future work ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Fort Saskatchewan Community Hospital, Ft Saskatchewan, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Since this is a pilot study we have no plans to share IPD with other researchers

REFERENCES:
- [Background] HerniaSurge Group. International guidelines for groin hernia management. Hernia. 2018 Feb;22(1):1-165. doi: 10.1007/s10029-017-1668-x. Epub 2018 Jan 12. PMID 29330835
- [Background] van Hanswijck de Jonge P, Lloyd A, Horsfall L, Tan R, O'Dwyer PJ. The measurement of chronic pain and health-related quality of life following inguinal hernia repair: a review of the literature. Hernia. 2008 Dec;12(6):561-9. doi: 10.1007/s10029-008-0412-y. Epub 2008 Aug 21. PMID 18716856
- [Background] Poobalan AS, Bruce J, Smith WC, King PM, Krukowski ZH, Chambers WA. A review of chronic pain after inguinal herniorrhaphy. Clin J Pain. 2003 Jan-Feb;19(1):48-54. doi: 10.1097/00002508-200301000-00006. PMID 12514456
- [Background] Cabilan CJ, Hines S, Munday J. The effectiveness of prehabilitation or preoperative exercise for surgical patients: a systematic review. JBI Database System Rev Implement Rep. 2015 Jan;13(1):146-87. doi: 10.11124/jbisrir-2015-1885. PMID 26447015
- [Background] Lundberg M, Archer KR, Larsson C, Rydwik E. Prehabilitation: The Emperor's New Clothes or a New Arena for Physical Therapists? Phys Ther. 2019 Feb 1;99(2):127-130. doi: 10.1093/ptj/pzy133. No abstract available. PMID 30508203
- [Background] Topp R, Ditmyer M, King K, Doherty K, Hornyak J 3rd. The effect of bed rest and potential of prehabilitation on patients in the intensive care unit. AACN Clin Issues. 2002 May;13(2):263-76. doi: 10.1097/00044067-200205000-00011. PMID 12011598
- [Background] Ditmyer MM, Topp R, Pifer M. Prehabilitation in preparation for orthopaedic surgery. Orthop Nurs. 2002 Sep-Oct;21(5):43-51; quiz 52-4. doi: 10.1097/00006416-200209000-00008. PMID 12432699
- [Background] Liang MK, Bernardi K, Holihan JL, Cherla DV, Escamilla R, Lew DF, Berger DH, Ko TC, Kao LS. Modifying Risks in Ventral Hernia Patients With Prehabilitation: A Randomized Controlled Trial. Ann Surg. 2018 Oct;268(4):674-680. doi: 10.1097/SLA.0000000000002961. PMID 30048306
- [Background] Nienhuijs SW, Rosman C, Strobbe LJ, Wolff A, Bleichrodt RP. An overview of the features influencing pain after inguinal hernia repair. Int J Surg. 2008 Aug;6(4):351-6. doi: 10.1016/j.ijsu.2008.02.005. Epub 2008 Mar 4. PMID 18450528
- [Background] Sobol-Kwapinska M, Babel P, Plotek W, Stelcer B. Psychological correlates of acute postsurgical pain: A systematic review and meta-analysis. Eur J Pain. 2016 Nov;20(10):1573-1586. doi: 10.1002/ejp.886. Epub 2016 May 2. PMID 27136510
- [Background] Schug SA, Lavand'homme P, Barke A, Korwisi B, Rief W, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic postsurgical or posttraumatic pain. Pain. 2019 Jan;160(1):45-52. doi: 10.1097/j.pain.0000000000001413. PMID 30586070
- [Background] Yeo AE, Berney CR. Carolinas Comfort Scale for mesh repair of inguinal hernia. ANZ J Surg. 2012 Apr;82(4):285-6. doi: 10.1111/j.1445-2197.2012.06012.x. No abstract available. PMID 22510195
- [Background] Heniford BT, Lincourt AE, Walters AL, Colavita PD, Belyansky I, Kercher KW, Sing RF, Augenstein VA. Carolinas Comfort Scale as a Measure of Hernia Repair Quality of Life: A Reappraisal Utilizing 3788 International Patients. Ann Surg. 2018 Jan;267(1):171-176. doi: 10.1097/SLA.0000000000002027. PMID 27655239
- [Derived] Shologan A, Farooq O, Bostick G, Macedo L, Durand-Moreau Q, Peters MR, Gross DP. A pilot randomized controlled trial examining the feasibility of perioperative rehabilitation for inguinal hernia repair surgery. PLoS One. 2025 May 22;20(5):e0324907. doi: 10.1371/journal.pone.0324907. eCollection 2025. PMID 40403095

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT05069142/Prot_SAP_ICF_000.pdf